CLINICAL TRIAL: NCT03465852
Title: HIV Prevention Among Latina Transgender Women Who Have Sex With Men: Evaluation of a Locally Developed Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00040441
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: The intervention study uses an intervention arm and a wait list comparison (control) arm
Who Masked: Outcomes Assessor
Masking Description: Study participants will be randomly assigned to the intervention or the wait list comparison arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Persons randomized to this arm will have completed the study consent process (including being tested with the INSTI rapid HIV test to verify their self-reported HIV negative status and their eligibility to participate in the study) and the baseline survey, and will receive the Spanish language ChiCAS intervention shortly after being randomized and will complete a follow-up assessment 6 months after completing the intervention.
  .
  Interventions: Behavioral: ChiCAS
- Wait list comparison (control) arm (Other): Persons randomized to this arm will have completed the study consent process (including being tested with the INSTI rapid HIV test to verify their self-reported HIV negative status and their eligibility to participate in the study) and the baseline survey, but will not receive the Spanish language ChiCAS intervention until they complete a follow-up assessment 6 months after completing the baseline assessment.
  Interventions: Behavioral: ChiCAS

INTERVENTIONS:
Behavioral: ChiCAS — Promotes access to and participation by HIV negative Hispanic/Latina transgender women who have sex with men in PrEP, medically supervised hormone therapy, and consistent condom use.

SUMMARY:
Wake Forest University and its partners, Triad Health Project, and the University of North Carolina, Greensboro, will be evaluating the effectiveness of ChiCAS (Chicas Creando Acceso a la Salud or Girls Creating Access to Health), a locally developed, Spanish language small group behavioral intervention that promotes access to and participation by Hispanic/Latina transgender women who are HIV negative and who have sex with men in pre-exposure prophylaxis (PrEP), medically supervised hormone therapy, and consistent condom use.

DETAILED DESCRIPTION:
ChiCAS will be delivered as two 4-hour group sessions over a period of two weeks to groups of about 10 participants at seven community-based organizations (CBOs) in five metropolitan locations in North Carolina (Asheville, Charlotte, Greensboro/Winston-Salem, Raleigh/Durham and Wilmington).

The intervention will be evaluated by comparing women randomized to the ChiCAS intervention group to those randomized to the delayed-intervention (waitlist) comparison group. As many as 140 participants (as many 70 participants per arm) in total will be recruited to the study. All participants will complete identical quantitative assessments at baseline and 6-month follow up. Baseline and 6-month follow-up data collection will include the following measures:

Outcome variables:

Use of PrEP and medically supervised hormone therapy and consistent condom use.

Demographics:

Age, current living situation, marital/partner status, education, country and region of origin, ethnicity/race, work and work patterns and history, financial status (including income, numbers of persons income supports), number of children and adults living in household, gender identity; time in the US and NC; Spanish-language literacy; English-language skills; health insurance; documentation status.

Mediating variables:

Knowledge about HIV and STDs: types of diseases, modes of transmission, signs, symptoms, prevention strategies, and their magnitude within communities; condom use-related attitudes, skills, self-efficacy, and intentions; adherence to traditional Latino values of masculinity and fatalism; transphobia; ethnic group pride; knowledge of available transition-related services, how to access, what to expect, and eligibility; barriers to seeking healthcare services, for HIV testing, PrEP, or transition-related services; perceived access to health care; social support; substance use; substance use during sex; communication skills with partners and providers; provider trust.

Other variables:

Religiosity; mental health, perceived discrimination; community attachment; foregoing unsafe sex/episodic abstinence HIV and sexually transmitted disease (STD) history; victimization; sexual compulsivity; sex for money, drugs or shelter, self-reported health status, acculturation, community attachment, technology use, HIV and STD history

A qualitative interview will be administered to 30 randomly selected participants after they complete the 6-month follow-up assessments. Three groups of ten participants each will be interviewed to identify factors associated with each of the following outcome patterns:

1. Participants who reported an increase in at least one HIV prevention behavioral outcome (PrEP or condom use) and who reported an increase in the use of medically supervised hormone therapy (n=10);
2. Participants who did not report an increase in at least one HIV prevention behavioral outcome (PrEP or condom use) and did not report an increase in the use of medically supervised hormone therapy (n=10), and
3. Participants with mixed results (n=10).

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify as male-to-female transgender or report having been born male and identifying as female;
2. Self-identify as Hispanic or Latina;
3. Are ≥ 18 years of age;
4. Report sex with at least 1 man in the past 6 months;
5. Are HIV negative (based on self-report and verification by HIV testing);
6. Are fluent in Spanish; and
7. Provide informed consent.

Exclusion Criteria:

(a) Having participated in any HIV prevention intervention within the past 12 months, including Chicas or other interventions co-developed by Wake Gorest University (HOLA en Grupos or HOLA).

* Are ≥ 18 years of age;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Persons who self-identify as male-to-female transgender or report having been born male and identifying as female.
Enrollment: 144 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Uptake of PrEP | Uptake compared to baseline assessed 6 months after completion of the intervention.
  Increased uptake of PrEP relative to baseline measures of use
Uptake of medically supervised hormone therapy | Uptake compared to baseline assessed 6 months after completion of the intervention.
  Increased uptake of medically supervised hormone therapy relative to baseline use measures
Consistent condom use | Uptake compared to baseline assessed 6 months after completion of the intervention.
  Increased consistent condom relative to baseline use measures

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Rhodes, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A plan agreed to by the Principal Investigator and the Centers for Disease Control and Prevention (CDC) will make, after approval by the CDC, the following study data available to applicants who provide detailed information on their reasons for requesting the data and plans analysis and use of the data:
  1. Quantitative data from structured surveys for baseline and 6-month follow-up assessments;
  2. Qualitative data from in-depth interviews with selected study participants to elucidate factors that contribute to or impede participant reports of engaging in the expected intervention outcomes following completion of the intervention (consistent condom use and use of PrEP and medically-supervised hormone therapy):
  3. medical record abstractions, and data from biological markers including PrEP and HIV test results. None of the data described here will contain personal identifying information from study participants.
Supporting Information: Study Protocol, SAP
Time Frame: Wake Forest University will make study data from which all personal identifying information has been removed, available to CDC for potential release at the termination of the study. It is anticipated that the complete dataset will be made available to CDC about April 2023, after the grantee, its partners, and CDC have agreed that all key study analyses have been completed and cleared by CDC for publication. All data will be retained until analysis is complete and for up to three years following study closure by the Wake Forest Institutional Review Board (IRB). At that time, users must delete all data stored on their servers. CDC will store complete de-identified data on a secure server that is accessible through the Division of HIV Prevention, Prevention Research Branch for an indefinite period.
Access Criteria: Persons who request data will be required to provide an approved copy of the Publication Guidelines Concept Proposal and a signed copy of the Data Sharing Agreement before data will be provided to them. The data sharing agreement must list and be signed by all individuals who will have access to the data or participate in preparing materials for publication before engaging in research and analysis activities with these data.